CLINICAL TRIAL: NCT00891085
Title: Synchronized Intermittent Mechanical Ventilation vs Open Lung Ventilation With Spontaneous Respiration
Brief Title: Synchronized Intermittent Mechanical Ventilation Versus Open Lung Ventilation With Spontaneous Respiration
Acronym: SOLV
Status: Terminated | Type: Observational
Why Stopped: unable to enroll patients adequately
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Jonathan Marinaro, professor, University of New Mexico
Other Study IDs: 07-302
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Last update posted 2023-05-19 (Actual); Status verified 2009-04

CONDITIONS: Trauma
Keywords: ventilation; ards; ali; trauma; Trauma Patients with ISS > 25
MeSH Terms: conditions — Wounds and Injuries; Respiratory Aspiration; Acute Lung Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Open Lung Ventilation: within 24 hours of arrival trauma patients with ISS >25 will be randomized to BiVent (APRV)
- SIMV: within 24 hours of arrival trauma patients with ISS >25 will be randomized to either SIMV or BiVent

SUMMARY:
The purpose of this study is to collect data on patients who are on breathing machines (ventilators) in the Trauma Surgical Intensive Care Unit (TSICU). This data may help us to determine if one form of assisted breathing is better than another. The two forms of assisted breathing being compared in this study are called BiVent and SIMV. (7) BiVent and SIMV are both delivered by a ventilator but differ in how they assist breathing. SIMV is an older form of mechanical breathing that blows air into the lungs to inflate the lungs. BiVent is a newer form of mechanical ventilation that permits the patient to pull air into the lungs as we normally do. Both BiVent and SIMV are currently being used on a regular basis in the TSICU. The investigators hope that this study will determine if one method of assisted breathing is better than another in preventing complications associated with mechanically assisted breathing.

DETAILED DESCRIPTION:
SOLV Hypothesis:

A prospective, randomized trial directly comparing open lung ventilation (OLV) with spontaneous breathing (SB) utilizing BiVent on the Maquet Servo-I versus synchronized intermittent mechanical ventilation (SIMV) will be conducted in the trauma-surgical intensive care unit at the University Hospital (TSICU). Both OLV-SB and SIMV protocols have been designed according to lung protective strategies. The primary goal of the SOLV trial is to see determine if the early application of open lung ventilation will less ventilator days. In addition, several secondary endpoints will be evaluated. It is not anticipated that this study will be powered to show a mortality difference.

ELIGIBILITY:
Inclusion Criteria:

* >/=18 years of age, ISS >/=25, on ventilator for more than 48 hours

Exclusion Criteria:

* less than 18 years of age, die or come off ventilator in less than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Trauma Patients with ISS>/=25
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Reduction in ventilator days | 4 years

SECONDARY OUTCOMES:
Progression to acute lung injury/acute respiratory distress syndrome (ALI/ARDS) | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States